CLINICAL TRIAL: NCT06658873
Title: Comparison of Proximal and Distal Cannulation of the Radial Artery by Ultrasonography in Adult Patients Undergoing Elective Surgery
Brief Title: Proximal vs Distal Radial Artery Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ruslan Abdullayev, Assoc. Prof. Dr., Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 09.2024.653
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Arterial Catheterization; Radial Artery Cannulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group P (Active Comparator): Radial arterial cannulation from the proximal part of the artery 5 cm proximal to the level of the styloid process.
  Interventions: Other: Proximal arterial cannulation
- Group D (Active Comparator): Radial arterial cannulation from the distal part of the artery at the styloid process.
  Interventions: Other: Distal arterial cannulation

INTERVENTIONS:
Other: Proximal arterial cannulation — Radial arterial cannulation from the proximal part of the artery 5 cm proximal to the level of the styloid process.
  Arms: Group P
Other: Distal arterial cannulation — Radial arterial cannulation from the distal part of the artery at the styloid process.
  Arms: Group D

SUMMARY:
Intraarterial cannulation is important for continuous blood pressure monitoring and blood gas analysis throughout the surgical procedure and in intensive care patients. Ultrasonography (USG) has gained popularity in vascular cannulations and facilitates intraarterial interventions. Radial artery is one of the most preferred arteries. Our aim in this study is to compare proximal and distal radial artery cannulations by USG in terms of procedural success, procedure time and complications.

DETAILED DESCRIPTION:
After the patients are admitted to the operating room, routine monitoring (electrocardiography, noninvasive blood pressure and peripheral oxygen saturation) will be performed. After appropriate vascular access is provided to the patients, the induction phase of general anesthesia will begin. Anesthesia induction will be left to the choice of the primary anesthesiologist and no protocol will be followed. In case of >25% drop in blood pressure, 0.1 mcg/kg noradrenaline will be administered intravenously. After the appropriate position is given to the arm of the patient to be treated, radial artery cannulation will be performed with USG obeying asepsis rules. Patients will be divided into 2 groups by closed envelope method. The first group will be the patients who will be cannulated at the level of the distal radius (styloid process) and the second group will be the patients who will be cannulated proximally by measuring 5 cm from the styloid process. Demographic and clinical characteristics of the patients will be recorded. Catheterization success rates, procedure duration, number of interventions, vessel diameter, hematoma at the site of intervention on the 1st postoperative day, circulatory disturbance will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* American Society of Anaesthesiologists (ASA) physical status I-III

Exclusion Criteria:

* Emergency surgery
* ASA IV or above
* Peripheral vascular disease
* Vasopressor use
* Anatomical abnormality at the cannulation site
* Infection at the cannulation site
* Coagulation defect

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Success | From the preinduction period in the operating theater to the postoperative day one.
  Radial artery catheterization success rates will be compared between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ruslan Abdullayev, Principal Investigator — Marmara University Department of Anesthesiology and Reanimation
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided